CLINICAL TRIAL: NCT00274430
Title: A Randomized Controlled Trial of the Effects of Tadalafil and Dexamethasone Versus Placebo on Pulmonary Edema Formation and Cerebral Blood Flow Autoregulation in High Altitude Newcomers With a Previous History of High Altitude Pulmonary Edema
Brief Title: Prevention of High Altitude Pulmonary Edema
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: margherita03
Record Dates: First submitted 2006-01-09; First posted 2006-01-10 (Estimated); Last update posted 2006-12-04 (Estimated); Status verified 2003-12

CONDITIONS: High Altitude Pulmonary Edema
MeSH Terms: conditions — Altitude Sickness | interventions — Dexamethasone; BID protein, human; Tadalafil

INTERVENTIONS:
Drug: dexamethasone 8 mg bid
Drug: tadalafil 10mg bid

SUMMARY:
A double-blind placebo controlled study

* To compare the effect of tadalafil and dexamethasone versus placebo on Ppa and pulmonary edema formation in subjects susceptible to HAPE.
* To investigate the effect of dexamethasone on alveolar fluid clearance, as assessed by measurement of the nasal potential difference, and prevention of HAPE.
* To investigate the effect of the tadalafil and dexamethasone versus placebo on the dynamic CBF autoregulation properties and on the development of AMS in HAPE susceptible subjects.

ELIGIBILITY:
Inclusion Criteria:

* At least one previous episode of high altitude pulmonary edema

Exclusion Criteria:

* pulmonary arterial hypertension
* congenital heart disease
* any chronic lung disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30
Dates: Start 2003-07; Study Completion 2003-09

PRIMARY OUTCOMES:
prevention of high altitude pulmonary edema

SECONDARY OUTCOMES:
incidence of acute mountain sickness

CONTACTS AND LOCATIONS:
Overall Officials: Marco Maggiorini, MD, Principal Investigator — University of Zurich

REFERENCES:
- [Result] Maggiorini M, Brunner-La Rocca HP, Peth S, Fischler M, Bohm T, Bernheim A, Kiencke S, Bloch KE, Dehnert C, Naeije R, Lehmann T, Bartsch P, Mairbaurl H. Both tadalafil and dexamethasone may reduce the incidence of high-altitude pulmonary edema: a randomized trial. Ann Intern Med. 2006 Oct 3;145(7):497-506. doi: 10.7326/0003-4819-145-7-200610030-00007. PMID 17015867
- [Derived] Clarenbach CF, Senn O, Christ AL, Fischler M, Maggiorini M, Bloch KE. Lung function and breathing pattern in subjects developing high altitude pulmonary edema. PLoS One. 2012;7(7):e41188. doi: 10.1371/journal.pone.0041188. Epub 2012 Jul 19. PMID 22829927